CLINICAL TRIAL: NCT04010214
Title: A Registered Cohort Study on Cerebellar Ataxia
Brief Title: A Registered Cohort Study on Cerebellar Ataxia in the Organization in South-East China for Cerebellar Ataxia Research (OSCCAR)
Status: Recruiting | Type: Observational
Sponsor: Ning Wang, MD., PhD. (Other)
Responsible Party: Sponsor-Investigator, Ning Wang, MD., PhD., The Vice President, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Other Study IDs: MRCTA,ECFAH of FMU[2019]195
Record Dates: First submitted 2019-07-04; First posted 2019-07-08 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Cerebellar Ataxia
MeSH Terms: conditions — Cerebellar Ataxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Cerebellar ataxia is a form of ataxia originating in the cerebellum. Cerebellar ataxia can occur as a result of many diseases and may present with symptoms of an inability to coordinate balance, gait, extremity and eye movements. To understand the clinical and genetic characteristics of cerebellar ataxia, we establish a registered cohort to follow up Chinese patients with cerebellar ataxia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cerebellar ataxia based on the diagnoses of tow neurologists
* Relatives of patients with cerebellar ataxia
* Unrelated healthy controls
* Participants or legal guardian(s) willing and able to complete the informed consent process

Exclusion Criteria:

* Participants are unable to comply with trial procedures and visit schedule

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cerebellar ataxia who are diagnosed by tow neurologists in the Organization in South-East China for Cerebellar Ataxia Research (OSCCAR) from the First Affiliated Hospital of Fujian Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2039-12 (Estimated); Study Completion 2059-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of hereditary cerebellar ataxia | Up to 20years
  Look for the causative gene in the patient with cerebellar ataxia

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology ,First Affiliated Hospital Fujian Medical University, Fuzhou, Fujian, China